CLINICAL TRIAL: NCT00440687
Title: Phase 4 Withdrawal of Inhaled Corticosteroids in Patients With Chronic Obstructive Pulmonary Disease in Primary Care: a Randomised Controlled Trial
Brief Title: Withdrawal of Inhaled Corticosteroids in Patients With COPD in Primary Care
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: British Lung Foundation (Other); GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QMUL - WISP 01; British Lung Foundation P00/8
Record Dates: First submitted 2007-02-26; First posted 2007-02-27 (Estimated); Last update posted 2007-02-27 (Estimated); Status verified 2007-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease; primary care; randomised trials; therapeutic interventions
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Fluticasone 500mcg BD via accuhaler or identical placebo

SUMMARY:
Guidelines recommend inhaled corticosteroids (ICS) for patients with moderate to severe chronic obstructive pulmonary disease (COPD). Most COPD patients are managed in primary care and receive ICS long-term and irrespective of severity. The effect of withdrawing ICS from COPD patients in primary care is unknown.This randomised double-blind placebo-controlled trial will evaluate the effect of withdrawal of inhaled corticosteroids in patients with COPD recruited from general practice. Participants will have a clinical and spirometric diagnosis of COPD and will have been prescribed inhaled steroids for the 6 months before entry to the trial. They will be randomised to taking a fixed dose steroid inhaler (Flixotide Accuhaler) or an identical placebo inhaler. Patients will be monitored using diary cards for a year with 3 monthly follow-up visits at their general practice. The primary outcome measures will be exacerbation frequency and severity. Other outcomes are time to first exacerbation, costs, health status, lung function and unscheduled care. We tested the hypothesis that withdrawal of ICS in this population would lead to an increased number of exacerbations, earlier onset of exacerbation, and a worsening of symptoms.

DETAILED DESCRIPTION:
To determine whether withdrawal of inhaled corticosteroids in patients with COPD in general practice effects:

* the frequency of exacerbations compared to a control group
* differences in health status compared to a control group
* differences in lung function compared to a control group
* changes in unscheduled care compared to a control group
* Direct and indirect costs compared to a control group

Hypothesis

The withdrawal of inhaled corticosteroids from patients with COPD identified in primary care will cause an increase in frequency and severity of exacerbations and is not cost-effective.

ELIGIBILITY:
Inclusion Criteria:

* Smoker or ex smoker of at least 10 pack years
* Age 40 or above
* Prior and current use of inhaled corticosteroids for at least 6 months duration (Used for at least 75% of time on direct questioning)
* FEV1 <80% of predicted, FEV1/FVC ratio <70%.
* Less than 15% change and <200 mls change in FEV1 20 minutes after 5 mg nebulised salbutamol.
* 256 patients to be included in trial of which 196 must have had a precious exacerbation of COPD in the last year

Exclusion Criteria:

* Clear history of asthma, bronchiectasis, carcinoma of bronchus or other significant respiratory disease
* Inability to give informed consent (severe mental illness, mental handicap or brain damage).
* Recorded exacerbation within last month that has required antibiotics or steroids (delayed randomisation)
* Classification as a never smoker
* Strongly positive skin allergy result (>10mm skin weal greater then negative control) to house dust mite, grass, tree, aspergillus, cat, dog or weed (irrespective of asthma/atopy status)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256
Dates: Start 2001-01; Study Completion 2004-03

PRIMARY OUTCOMES:
the frequency of exacerbations compared to a control group

SECONDARY OUTCOMES:
differences in time to first exacerbation compared to control group
differences in health status compared to a control group
differences in lung function compared to a control group
changes in unscheduled care compared to a control group
direct and indirect costs compared to a control group
comparison of side effects between groups

CONTACTS AND LOCATIONS:
Overall Officials: Aklak B Choudhury, MRCP, Principal Investigator — Centre for Health Sciences, Queen Mary's School of Medicine and Dentistry; Gene S Feder, MRCGP MD, Study Chair — Centre for Health Sciences, Queen Mary's School of Medicine and Dentistry; Jadwiga A Wedzicha, MRCP MD, Study Chair — Academic Unit of Respiratory Medicine, Royal Free and University College Medical School; Chris J Griffiths, MRCP MRCGP MD, Study Director — Centre for Health Sciences, Queen Mary's School of Medicine and Dentistry
Locations (1):
- Centre for Health Sciences, Queen Mary's School of Medicine and Dentistry, Barts and The London, 2 Newark Street,., London and Essex, London, United Kingdom

REFERENCES:
- [Background] Seemungal TA, Donaldson GC, Paul EA, Bestall JC, Jeffries DJ, Wedzicha JA. Effect of exacerbation on quality of life in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 1998 May;157(5 Pt 1):1418-22. doi: 10.1164/ajrccm.157.5.9709032. PMID 9603117
- [Background] Miravitlles M, Ferrer M, Pont A, Zalacain R, Alvarez-Sala JL, Masa F, Verea H, Murio C, Ros F, Vidal R; IMPAC Study Group. Effect of exacerbations on quality of life in patients with chronic obstructive pulmonary disease: a 2 year follow up study. Thorax. 2004 May;59(5):387-95. doi: 10.1136/thx.2003.008730. PMID 15115864
- [Background] McGuire A, Irwin DE, Fenn P, Gray A, Anderson P, Lovering A, MacGowan A. The excess cost of acute exacerbations of chronic bronchitis in patients aged 45 and older in England and Wales. Value Health. 2001 Sep-Oct;4(5):370-5. doi: 10.1046/j.1524-4733.2001.45049.x. PMID 11705127
- [Background] Davies L, Angus RM, Calverley PM. Oral corticosteroids in patients admitted to hospital with exacerbations of chronic obstructive pulmonary disease: a prospective randomised controlled trial. Lancet. 1999 Aug 7;354(9177):456-60. doi: 10.1016/s0140-6736(98)11326-0. PMID 10465169
- [Background] Donaldson GC, Seemungal TA, Bhowmik A, Wedzicha JA. Relationship between exacerbation frequency and lung function decline in chronic obstructive pulmonary disease. Thorax. 2002 Oct;57(10):847-52. doi: 10.1136/thorax.57.10.847. PMID 12324669
- [Background] Kanner RE, Anthonisen NR, Connett JE; Lung Health Study Research Group. Lower respiratory illnesses promote FEV(1) decline in current smokers but not ex-smokers with mild chronic obstructive pulmonary disease: results from the lung health study. Am J Respir Crit Care Med. 2001 Aug 1;164(3):358-64. doi: 10.1164/ajrccm.164.3.2010017. PMID 11500333
- [Background] Spencer S, Calverley PM, Burge PS, Jones PW. Impact of preventing exacerbations on deterioration of health status in COPD. Eur Respir J. 2004 May;23(5):698-702. doi: 10.1183/09031936.04.00121404. PMID 15176682
- [Background] Burge PS, Calverley PM, Jones PW, Spencer S, Anderson JA, Maslen TK. Randomised, double blind, placebo controlled study of fluticasone propionate in patients with moderate to severe chronic obstructive pulmonary disease: the ISOLDE trial. BMJ. 2000 May 13;320(7245):1297-303. doi: 10.1136/bmj.320.7245.1297. PMID 10807619
- [Background] Calverley P, Pauwels R, Vestbo J, Jones P, Pride N, Gulsvik A, Anderson J, Maden C; TRial of Inhaled STeroids ANd long-acting beta2 agonists study group. Combined salmeterol and fluticasone in the treatment of chronic obstructive pulmonary disease: a randomised controlled trial. Lancet. 2003 Feb 8;361(9356):449-56. doi: 10.1016/S0140-6736(03)12459-2. PMID 12583942
- [Background] Paggiaro PL, Dahle R, Bakran I, Frith L, Hollingworth K, Efthimiou J. Multicentre randomised placebo-controlled trial of inhaled fluticasone propionate in patients with chronic obstructive pulmonary disease. International COPD Study Group. Lancet. 1998 Mar 14;351(9105):773-80. doi: 10.1016/s0140-6736(97)03471-5. PMID 9519948
- [Background] Alsaeedi A, Sin DD, McAlister FA. The effects of inhaled corticosteroids in chronic obstructive pulmonary disease: a systematic review of randomized placebo-controlled trials. Am J Med. 2002 Jul;113(1):59-65. doi: 10.1016/s0002-9343(02)01143-9. PMID 12106623
- [Background] National Collaborating Centre for Chronic Conditions. Chronic obstructive pulmonary disease. National clinical guideline on management of chronic obstructive pulmonary disease in adults in primary and secondary care. Thorax. 2004 Feb;59 Suppl 1(Suppl 1):1-232. No abstract available. PMID 15041752
- [Background] Pauwels RA, Buist AS, Calverley PM, Jenkins CR, Hurd SS; GOLD Scientific Committee. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease. NHLBI/WHO Global Initiative for Chronic Obstructive Lung Disease (GOLD) Workshop summary. Am J Respir Crit Care Med. 2001 Apr;163(5):1256-76. doi: 10.1164/ajrccm.163.5.2101039. No abstract available. PMID 11316667
- [Background] Herland K, Akselsen JP, Skjonsberg OH, Bjermer L. How representative are clinical study patients with asthma or COPD for a larger "real life" population of patients with obstructive lung disease? Respir Med. 2005 Jan;99(1):11-9. doi: 10.1016/j.rmed.2004.03.026. PMID 15672843
- [Background] Tirimanna PR, van Schayck CP, den Otter JJ, van Weel C, van Herwaarden CL, van den Boom G, van Grunsven PM, van den Bosch WJ. Prevalence of asthma and COPD in general practice in 1992: has it changed since 1977? Br J Gen Pract. 1996 May;46(406):277-81. PMID 8762742
- [Background] van Schayck CP, Levy ML, Stephenson P, Sheikh A. The IPCRG Guidelines: developing guidelines for managing chronic respiratory diseases in primary care. Prim Care Respir J. 2006 Feb;15(1):1-4. doi: 10.1016/j.pcrj.2005.12.003. Epub 2006 Jan 18. No abstract available. PMID 16701751
- [Background] Seemungal TA, Donaldson GC, Bhowmik A, Jeffries DJ, Wedzicha JA. Time course and recovery of exacerbations in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2000 May;161(5):1608-13. doi: 10.1164/ajrccm.161.5.9908022. PMID 10806163
- [Background] Anthonisen NR, Manfreda J, Warren CP, Hershfield ES, Harding GK, Nelson NA. Antibiotic therapy in exacerbations of chronic obstructive pulmonary disease. Ann Intern Med. 1987 Feb;106(2):196-204. doi: 10.7326/0003-4819-106-2-196. PMID 3492164
- [Background] Jones PW, Quirk FH, Baveystock CM, Littlejohns P. A self-complete measure of health status for chronic airflow limitation. The St. George's Respiratory Questionnaire. Am Rev Respir Dis. 1992 Jun;145(6):1321-7. doi: 10.1164/ajrccm/145.6.1321. PMID 1595997
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Vestbo J, Sorensen T, Lange P, Brix A, Torre P, Viskum K. Long-term effect of inhaled budesonide in mild and moderate chronic obstructive pulmonary disease: a randomised controlled trial. Lancet. 1999 May 29;353(9167):1819-23. doi: 10.1016/s0140-6736(98)10019-3. PMID 10359405
- [Background] Wouters EF, Postma DS, Fokkens B, Hop WC, Prins J, Kuipers AF, Pasma HR, Hensing CA, Creutzberg EC; COSMIC (COPD and Seretide: a Multi-Center Intervention and Characterization) Study Group. Withdrawal of fluticasone propionate from combined salmeterol/fluticasone treatment in patients with COPD causes immediate and sustained disease deterioration: a randomised controlled trial. Thorax. 2005 Jun;60(6):480-7. doi: 10.1136/thx.2004.034280. PMID 15923248
- [Background] van der Valk P, Monninkhof E, van der Palen J, Zielhuis G, van Herwaarden C. Effect of discontinuation of inhaled corticosteroids in patients with chronic obstructive pulmonary disease: the COPE study. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1358-63. doi: 10.1164/rccm.200206-512OC. Epub 2002 Sep 5. PMID 12406823
- [Background] O'Brien A, Russo-Magno P, Karki A, Hiranniramol S, Hardin M, Kaszuba M, Sherman C, Rounds S. Effects of withdrawal of inhaled steroids in men with severe irreversible airflow obstruction. Am J Respir Crit Care Med. 2001 Aug 1;164(3):365-71. doi: 10.1164/ajrccm.164.3.2002052. PMID 11500334
- [Background] Jarad NA, Wedzicha JA, Burge PS, Calverley PM. An observational study of inhaled corticosteroid withdrawal in stable chronic obstructive pulmonary disease. ISOLDE Study Group. Respir Med. 1999 Mar;93(3):161-6. doi: 10.1016/s0954-6111(99)90001-x. PMID 10464871
- [Background] Jones PW, Willits LR, Burge PS, Calverley PM; Inhaled Steroids in Obstructive Lung Disease in Europe study investigators. Disease severity and the effect of fluticasone propionate on chronic obstructive pulmonary disease exacerbations. Eur Respir J. 2003 Jan;21(1):68-73. doi: 10.1183/09031936.03.00013303. PMID 12570111
- [Background] Pauwels RA, Lofdahl CG, Laitinen LA, Schouten JP, Postma DS, Pride NB, Ohlsson SV. Long-term treatment with inhaled budesonide in persons with mild chronic obstructive pulmonary disease who continue smoking. European Respiratory Society Study on Chronic Obstructive Pulmonary Disease. N Engl J Med. 1999 Jun 24;340(25):1948-53. doi: 10.1056/NEJM199906243402503. PMID 10379018
- [Derived] Choudhury AB, Dawson CM, Kilvington HE, Eldridge S, James WY, Wedzicha JA, Feder GS, Griffiths CJ. Withdrawal of inhaled corticosteroids in people with COPD in primary care: a randomised controlled trial. Respir Res. 2007 Dec 27;8(1):93. doi: 10.1186/1465-9921-8-93. PMID 18162137